CLINICAL TRIAL: NCT06157944
Title: Diagnostic Reasoning With Large Language Model Chat Bots
Brief Title: Physician Reasoning on Diagnostic Cases With Large Language Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Jonathan Chen, Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 71319
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Diagnosis
Keywords: Computer-assisted diagnosis; Large language models; clinical reasoning
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: The trial will be designed as a randomized, two-arm, single-blind parallel group study.
Who Masked: Outcomes Assessor
Masking Description: The grading of responses will be performed by assessors blinded to participant identity and treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPT-4 (Active Comparator): Group will be given access to GPT-4.
  Interventions: Other: GPT-4
- Usual resources (No Intervention): Group will not be given access to GPT-4 but will be encouraged to use any resources they wish besides large language models (UpToDate, Dynamed, google, etc).

INTERVENTIONS:
Other: GPT-4 — OpenAI's GPT-4 large language model with chat interface.
  Arms: GPT-4

SUMMARY:
This study will evaluate the effect of providing access to GPT-4, a large language model, compared to traditional diagnostic decision support tools on performance on case-based diagnostic reasoning tasks.

DETAILED DESCRIPTION:
Artificial intelligence (AI) technologies, specifically advanced large language models like OpenAI's ChatGPT, have the potential to improve medical decision-making. Although ChatGPT-4 was not developed for its use in medical-specific applications, it has demonstrated promise in various healthcare contexts, including medical note-writing, addressing patient inquiries, and facilitating medical consultation. However, little is known about how ChatGPT augments the clinical reasoning abilities of clinicians.

Clinical reasoning is a complex process involving pattern recognition, knowledge application, and probabilistic reasoning. Integrating AI tools like ChatGPT-4 into physician workflows could potentially help reduce clinician workload and decrease the likelihood of missed diagnoses. However, ChatGPT-4 was not developed for the purpose of clinical reasoning nor has it been validated for this purpose. Further, it may be subject to disinformation, including convincing confabulations that may mislead clinicians. If clinicians misuse this tool, it may not improve diagnostic reasoning and could even cause harm. Therefore, it is important to study how clinicians use large language models to augment clinical reasoning prior to routine incorporation into patient care.

In this study, we will randomize participants to answer diagnostic cases with or without access to ChatGPT-4. The participants will be asked to give three differential diagnoses for each case, with supporting and opposing findings for each diagnosis. Additionally they will be asked to provide their top diagnosis along with next diagnostic steps. Answers will be graded by independent reviewers blinded to treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be licensed physicians and have completed at least post-graduate year 2 (PGY2) of medical training.
* Training in Internal medicine, family medicine, or emergency medicine.

Exclusion Criteria:

* Not currently practicing clinically.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic reasoning | During evaluation
  The primary outcome will be the percent correct (range: 0 to 100) for each case. For each case, participants will be asked for three top diagnoses and findings from the case that support that diagnosis and oppose that diagnosis. Participants will receive 1 point for each plausible diagnosis. Findings supporting the diagnosis and findings opposing the diagnosis will also be graded based on correctness, with 1 point for partially correct and 2 points for completely correct responses. Participants will then be asked to name their top diagnosis, earning one point for a reasonable response and two points for the most correct response. Finally participants will be asked to name up to 3 next steps to further evaluate the patient with one point awarded for a partially correct response and two points for a completely correct response. The primary outcome will be compared on the case-level by the randomized groups.

SECONDARY OUTCOMES:
Time Spent on Diagnosis | During evaluation
  We will compare how much time (in minutes) participants spend per case between the two study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan H Chen, MD, PhD, Principal Investigator — Stanford University; Adam Rodman, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Andrew Olson, MD, Principal Investigator — University of Minnesota
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goh E, Gallo R, Hom J, Strong E, Weng Y, Kerman H, Cool JA, Kanjee Z, Parsons AS, Ahuja N, Horvitz E, Yang D, Milstein A, Olson APJ, Rodman A, Chen JH. Large Language Model Influence on Diagnostic Reasoning: A Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2440969. doi: 10.1001/jamanetworkopen.2024.40969. PMID 39466245